CLINICAL TRIAL: NCT02200237
Title: A Clinical Study for Inactivated Vaccine Against EV71
Acronym: EV71
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medigen Vaccine Biologics Corp. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CT-EV-21
Record Dates: First submitted 2014-07-18; First posted 2014-07-25 (Estimated); Last update posted 2017-08-18 (Actual); Status verified 2017-08

CONDITIONS: Enterovirus 71 Human
Keywords: EV71 Vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Phosphate Buffer Saline with adjuvant aluminium phosphate
  Interventions: Biological: Placebo
- EV71 with adjuvant aluminium phosphate (Experimental): Inactive whole monovalent EV71 virion vaccine formulated with phosphate-buffered saline based adjuvanted aluminium phosphate 150 μg/0.5ml
  Interventions: Biological: EV71 with adjuvant aluminium phosphate

INTERVENTIONS:
Biological: EV71 with adjuvant aluminium phosphate — Two arms, EV71 with aluminium phosphate
  Arms: EV71 with adjuvant aluminium phosphate
Biological: Placebo — Phosphate Buffer Saline with adjuvant aluminium phosphate
  Arms: Placebo

SUMMARY:
This study aims to evaluate the safety, reactogenicity and immunogenicity of EV71 vaccine in health children and infants aged from 2 months to <12yrs.

ELIGIBILITY:
Main Inclusion Criteria:

1. Healthy children and infants aged from 2 months to less than 12 years as established by medical history and clinical examination
2. The subjects' guardians are able to understand and sign the informed consent

Main Exclusion Criteria:

1. Subject with previous known exposure to EV71.
2. Subject with a history of herpangina or hand, foot and mouth disease associated with enterovirus infection in the past 3 months.
3. Subject who was diagnosed with a significant neurological, pulmonary, cardiovascular, hematological, hepatic or renal disorder.
4. Use of any investigational/non-registered product (including drug, vaccine and invasive medical device) within 30 days prior to vaccination or planned use during study period.
5. Subject with any confirmed or suspected autoimmune disorder, or immunodeficiency
6. Use of immunoglobulins or any blood products within 3 months prior to vaccination or planned use during the whole study period.

Ages: 2 Months to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 366 (Actual)
Dates: Start 2014-09; Primary Completion 2017-05 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
To evaluate overall safety of EV71 vaccine in children, throughout the study period | 2 years after study initiation
  Occurrence of overall adverse events and serious adverse events during the entire period of study.

SECONDARY OUTCOMES:
To evaluate immunogenicity, serum neutralizing antibody titers humoral immune response, induced by candidate vaccine | 2 years from study initiation
  To evaluate the immunogencity in terms of
  * Geometric mean titer (GMT) of EV71 neutralizing antibody titers
  * Post-vaccination-to-pre-vaccination GMT ratio of EV 71 neutralizing antibody titers
  * Seropositivity rate

CONTACTS AND LOCATIONS:
Overall Officials: Li-Min Huang, M.D., PhD., Principal Investigator — National Taiwan University Hospital
Locations (4):
- Taiwan (4):
  - Chang-Guang Memorial Hospital Lin-Kou, Taipei
  - Far Eastern Memorial Hospital, Taipei
  - MacKay Memorial Hospital, Taipei
  - National Taiwan University Hosptial, Taipei